CLINICAL TRIAL: NCT03622125
Title: Decrease in Temperature by Scorpion Sting: a Pagtonomic Sign
Brief Title: Decrease in Temperature as a Pagtonomic Sign by Scorpion Sting
Status: Completed | Type: Observational
Sponsor: Mexican Red Cross (Other)
Collaborators: Instituto Bioclon S.A. de C.V. (Industry)
Responsible Party: Principal Investigator, Josue Saul Almaraz Lira, Principal Investigator, Mexican Red Cross
Other Study IDs: CRM-Alacranes-2017
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-08

CONDITIONS: Scorpion Stings
MeSH Terms: conditions — Scorpion Stings | interventions — Vital Signs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients who apply anti-scorpion venom serum Birmex at the discretion of the attending physician were given vital signs.
  Interventions: Diagnostic Test: Vital signs
- 2: Patients who apply anti-scorpion venom serum Alacramyn at the discretion of the attending physician were given vital signs.
  Interventions: Diagnostic Test: Vital signs

INTERVENTIONS:
Diagnostic Test: Vital signs — Axillary temperature sampling, at the site of the scorpion sting and the contralateral site with infrared thermometer, and heart rate, respiratory rate and blood pressure on admission, 30 minutes after applying the vial and the medical discharge

SUMMARY:
The scorpion sting is a medical disease, for the signs and symptoms presented; Sometimes patients do not know the animal that causes these symptoms; the bibliography marks the decrease in temperature as a sign to be presented.

DETAILED DESCRIPTION:
The scorpion sting is a medical emergency where 184 patients from the state of Guanajuato were divided into 2 groups according to the type of antivenom administered, the dose of antivenom were at the discretion of the attending physician, Birmex (n = 117) and Alacramyn (n = 67) for the temperature record of the site of sting and other vital signs, this to compare it with the bibliography as a pathognomonic sign.

ELIGIBILITY:
Inclusion Criteria:

* Scorpion sting
* All sex
* 3 - 90 ages

Exclusion Criteria:

* Application of ice at the sting site

Ages: 3 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Person who has been scorpion sting and present signs and symptoms of poisoning to will applied a treatment in the city of León, Guanajuato
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Temperature change | 0, 30 and 120 minutes
  Temperature at the sting site, contralateral site and axillary in degrees celcius

SECONDARY OUTCOMES:
Blood preasure | 0, 30 and 120 minutes
  Systolic and diastolic in mmHg
Heart rate | 0, 30 and 120 minutes
  Beats per minute
Respiratory rate | 0, 30 and 120 minutes
  Breaths per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Cruz Roja Mexicana, Delegación León, León, Guanajuato, Mexico

REFERENCES:
- [Background] Isbister GK, Bawaskar HS. Scorpion envenomation. N Engl J Med. 2014 Jul 31;371(5):457-63. doi: 10.1056/NEJMra1401108. No abstract available. PMID 25075837